CLINICAL TRIAL: NCT00348257
Title: Safety and Efficacy of Using LEORTEC-300 System For Hair Removal Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leortec Medical Systems Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEORTC-HR-001
Record Dates: First submitted 2006-07-02; First posted 2006-07-04 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Epilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Hair removal by laser/IPL device

SUMMARY:
Removal of unwanted hair is one of the most commonly sought cosmetic solutions. Traditional methods, such as shaving, depilatories, tweezing and waxing result in only temporary hair removal, and thus require extensive maintenance. Long term hair removal via electrolysis is generally unsatisfactory due to its time consuming, painful nature and the associated risk of scarring or pigmentary changes. Moreover, the efficacy of electrolysis is user dependent and is estimated to be reduction of only 15-50% of the unwanted hair3.

The more modern approach to long term hair removal involves laser and Intense Pulsed Light (IPL) treatment modalities. These technologies are based on the scientific principle of selective photothermolysis. During the treatment, the light energy is absorbed by the hair's pigment (melanin) and transmitted through the hair shaft to the follicle. Conversion of this energy into heat causes a rise in the hair temperature, leading to destruction of the follicle and disruption of the hair growth mechanism, while leaving the skin undamaged.

Both laser and light devices have been proven successful in inducing permanent hair removal, as well as delayed hair growth, while causing minimal discomfort and complications. The light devices are based on the IPL technology, which differs from laser light in various physical aspects. The main difference is that while lasers emit light at a distinct wavelength, IPL delivers a wide range of wavelengths (400 1400 nm), thus allowing greater flexibility in aspects of body area, hair color and skin type LEORTEC LTD. has developed an innovative device that integrates the two treatment modalities: Laser and Intense Pulse Light (IPL) and in addition MLS - Multi Light Source- a combination of the two modalities. The purpose of this study is to evaluate the safety and efficacy of using Leortec 300 device for hair removal treatment.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

1. Primary Objective

   * Safety

     * To evaluate the safety of using LEORTEC-300 System for hair removal treatment, in different skin/hair colors and anatomical sites.
2. Secondary Objectives

   * Effectiveness

     * To assess the effectiveness of using the LEORTEC-300 system for hair removal treatment in different skin/hair colors and anatomical sites.
     * Patient Satisfaction Immediately after the treatment patients will be asked to rate pain level which they felt during the treatment.
     * Physician's Satisfaction Physician's satisfaction from the technique, equipment and hair removal will be assessed by physician's questionnaire.

STUDY DESIGN

This is a two-sites, prospective, controlled study to further test the safety and effectiveness of the LEORTEC-300 system in hair removal treatment.

SUBJECTS

1.Source and Number Subjects for the study will be recruited from patients within the community who have sought treatment for hair removal from the investigative physicians and meet all of the eligibility criteria listed below. There will be a total of 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males/females between the ages of 18 to 70
* Subject is willing to go trough hair removal treatment.
* Subject understands the study procedure.
* Subject is willing to sign the inform consent.
* Subject must have the ability to comply with the study procedures and follow- up.

Exclusion Criteria:

* Age < 18 years or > 70 years.
* Use of medication for which 400nm to 1400nm light exposure is contraindicated
* Coagulation disorder.
* Infection / abscess / pains in treatment target area.
* Recently tanned skin.
* Photosensitivity or allergy.
* Psoriasis.
* Skin cancer.
* Diabetes.
* Pregnancy.
* Tattoo on targeted area.
* History of keloid scarring.
* Use of aspirin or antioxidants
* Eczema or dermatitis.
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol.
* Physician objection.
* Known cognitive or psychiatric disorder
* Participation in any other clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-07; Study Completion 2006-09

PRIMARY OUTCOMES:
Hair removal efficiency 1- N1/N2 (N1 - Average number of hairs after the treatment
N2 - Average number of hairs before the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Levy, PhD, Study Director — Leortec Medical Systems
Locations (1):
- Elisha Hospital, Haifa, Israel